CLINICAL TRIAL: NCT02429856
Title: SCORPIO™ Posterior Stabilized Versus Posterior Retained Total Knee Arthroplasties: Long-term Functional and Radiographic Outcome
Brief Title: Posterior Cruciate Retaining (PCR) Versus Posterior Cruciate Substituting (PCS) Total Knee Arthroplasty (TKA)
Acronym: SCORPIO™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00002407
Record Dates: First submitted 2015-04-17; First posted 2015-04-29 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Arthroplasty, Replacement, Knee; Knee Arthroplasty, Total

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCS (Active Comparator): SCORPIO™ Posterior Cruciate Ligament Substituting TKA prosthesis
  Interventions: Device: SCORPIO™
- PCR (Active Comparator): SCORPIO™ Posterior Cruciate Ligament Retaining TKA prosthesis
  Interventions: Device: SCORPIO™

INTERVENTIONS:
Device: SCORPIO™ — subjects randomized at surgery to receive 1 of the 2 specified implants

SUMMARY:
This randomized clinical trial (RCT) examined 10 year outcomes comparing SCORPIO™ Posterior Cruciate Substituting (PCS) versus Posterior Cruciate Retaining (PCR) Total Knee Arthroplasty (TKA) as the primary outcome.

DETAILED DESCRIPTION:
RCT of 100 subjects undergoing primary TKA who were randomized to received either a SCORPIO™ PCS or PCR TKA.

Subjects were evaluated pre-operatively and at 2 and 10 years post-operatively using the Western Ontario (WOMAC) Osteoarthritis Index, the RAND-36 and knee range of motion (2 years only). Complication and revision rates were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for primary TKA
* non-inflammatory arthritis
* intact Posterior Cruciate Ligament at the time of surgery

Exclusion Criteria:

* required bone grafting of either the femur or tibia
* varus or valgus deformity of > 15 degrees
* previous high tibial osteotomy
* unable to understand or comply with the study requirements
* unable to provide signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 1999-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Health Services - Edmonton zone, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Chaudhary R, Beaupre LA, Johnston DW. Knee range of motion during the first two years after use of posterior cruciate-stabilizing or posterior cruciate-retaining total knee prostheses. A randomized clinical trial. J Bone Joint Surg Am. 2008 Dec;90(12):2579-86. doi: 10.2106/JBJS.G.00995. PMID 19047702

RESULTS

PARTICIPANT FLOW:
Groups:
- PCS Group: SCORPIO™ Posterior Cruciate Ligament Substituting TKA prosthesis
  SCORPIO™: subjects randomized at surgery to receive 1 of the 2 specified TKA implants
- PCR Group: SCORPIO™ Posterior Cruciate Ligament Retaining TKA prosthesis
  SCORPIO™: subjects randomized at surgery to receive 1 of the 2 specified implants
Period: Overall Study
Arm/Group | PCS Group | PCR Group
Started | 49 | 51
Completed | 30 | 32
Not Completed | 19 | 19
Not completed — Death | 12 | 13
Not completed — Lost to Follow-up | 6 | 5
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- PCS Group: SCORPIO™ Posterior Cruciate Ligament Substituting TKA prosthesis
  SCORPIO™: subjects randomized at surgery to receive 1 of the 2 specified implants
- Total: Total of all reporting groups
Arm/Group | PCS Group | PCR Group | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 49 | 51 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (8.4) | 69.2 (9.1) | 69.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 49
  Male | 27 | 24 | 51
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario McMaster (WOMAC) Osteoarthritis Index Pain
Description: disease-specific patient reported health related quality of life (pain and function) with 2 constructs (pain; function) each ranging from 0-100 points No total score is calculated; we report the WOMAC in reverse order to align with the RAND-36 scores where higher scores are considered better than lower scores
Time Frame: 10 years postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PCR Group: SCORPIO™ Posterior Cruciate Ligament Retaining TKA prosthesis
  SCORPIO™: subjects randomized at surgery to receive 1 of the 2 specified TKA implants
Arm/Group | PCS Group | PCR Group
Number analyzed (Participants) | 30 | 32
units on a scale | 84.0 (19.8) | 78.3 (24.5)

2. Primary Outcome: WOMAC Osteoarthritis Index Function
Description: as for outcome 1
Time Frame: 10 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PCS Group | PCR Group
Number analyzed (Participants) | 26 | 30
units on a scale | 67.9 (25.6) | 72.7 (23.3)

3. Secondary Outcome: RAND -36 Health Survey
Description: generic patient reported health related quality of life measure with 8 dimensions of health - we report the physical function dimension only with scores ranging from 0-100 where higher scores indicate better physical function.
Time Frame: 10 years postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PCS Group | PCR Group
Number analyzed (Participants) | 30 | 32
units on a scale | 42.4 (28.7) | 50.3 (29.3)

4. Secondary Outcome: Revision Rate
Description: number of participants with revision surgery (ie another surgery on the same knee) for any cause data obtained from patient report and regional administrative databases
Time Frame: within 10 years of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | PCS Group | PCR Group
Number analyzed (Participants) | 30 | 32
Participants | 5 | 2

5. Secondary Outcome: Number of Complications
Time Frame: within 10 years of surgery
Population: These complications include the revisions already recorded.
Measure: Count of Participants; unit: Participants
Arm/Group | PCS Group | PCR Group
Number analyzed (Participants) | 32 | 30
Participants | 6 | 2

6. Secondary Outcome: Knee Range of Motion
Description: Knee Range of Motion measured as a calculated total of knee flexion + knee extension; measured in degrees
Time Frame: knee ROM at 2 years postoperative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | PCS Group | PCR Group
Number analyzed (Participants) | 38 | 40
degrees | 105.8 (13.5) | 105.9 (13.0)

ADVERSE EVENTS:
Arm/Group | PCS Group | PCR Group
Serious Adverse Events (participants affected / at risk) | 5/49 | 2/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCS Group (N=49) | PCR Group (N=51)
Revision of TKA (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No